CLINICAL TRIAL: NCT03551938
Title: ATN 157 -We Prevent: A Dyadic Approach to HIV Prevention and Care Among Young Male Couples
Brief Title: We Prevent: A Dyadic Approach to HIV Prevention and Care Among Young Male Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: FWA00004801; 5U19HD089881-04 (NIH)
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: HIV/AIDS
Keywords: HIV, telehealth, HIV testing, YMSM, couples
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Family Characteristics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Receive only the standard HIV Counseling, Testing, and Referral or Couples HIV Testing and Counseling (CHTC) Session.
- Intervention (Experimental): Receive one 45-minute Relationship skills session for YMSM individuals and couples (the intervention) as an addition to the standard HIV Counseling, Testing, and Referral (CTR) or Couples HIV Testing and Counseling (CHTC) Session.
  Interventions: Behavioral: Relationship skills session for YMSM partnered-individuals and couples

INTERVENTIONS:
Behavioral: Relationship skills session for YMSM partnered-individuals and couples — Relationship skills session as an addition to the current CTR and CHTC intervention for 15-24 year old YMSM and their partners.
  Arms: Intervention

SUMMARY:
We Prevent seeks to develop and pilot test a developmentally-appropriate relationship skills session as an addition to the current Couples HIV Testing and Counseling (CHTC) intervention for young gay, bisexual and other men who have sex with men (YMSM). This project involves three phases to develop and pilot test the intervention. Phase I collected brief quantitative survey data, in-depth qualitative interview data, and cognitive interview data from YMSM and feedback from a technical expert group (TEG) to develop and refine the two-session intervention. Phase II involved conducting a one-arm pilot of the intervention condition to further refine the intervention content with a sample of 12 YMSM (6 dyads). Phase III involves conducting a randomized controlled trial (RCT) comparing the relationship-focused intervention to a control condition, which is HIV Testing, Counseling, and Referrals (CTR) alone with a sample of 320 YMSM.

DETAILED DESCRIPTION:
Young (15-24 years old) gay, bisexual and other men who have sex with men (YMSM) continue to be the group most heavily impacted by HIV in the US, despite stable or declining rates of infection among other groups. HIV prevention and research efforts in the US have continued to target MSM as individuals, largely focusing on messages that encourage the uptake of prevention efforts and reducing sexual risk. Recently, there has been growing interest in structural interventions to reduce HIV risk, tackling social, economic and cultural factors that place MSM in contexts of risk. However, despite socio-ecological theory postulating the importance of individual, dyadic and social influences on HIV risk, there has been a dearth of intervention efforts focused at the dyadic level.

We Prevent seeks to intervene on relationship communication skills as a pathway to HIV prevention during the critical period of adolescence. The proposed activities will develop and test a relationship skills focused HIV prevention intervention for young YMSM aged 15-24 as an addition to the current HIV Counseling, Testing, and Referrals (CTR) and Couples HIV Testing and Counseling (CHTC). At home STI test kits will also be sent in Phases II and III at baseline and one follow up.

Phase I of the project included collection of data from two groups of participants: 1) 30 YMSM in in-depth interviews and 8 YMSM in cognitive interviews and 2) 7 Technical Experts (TEG), for a total sample of 45 research participants.

Phase II consisted of a one-arm pilot test of the intervention condition with 6 YMSM dyads (total 12 participants). Participants completed a Baseline and 1-month follow-up assessment.

Phase III involves a pilot two-arm prospective RCT in which 320 YMSM will complete a Baseline assessment and then complete assessments every 3 months for 9 months.

Recruitment of all participants is in all 50 states and will be conducted through popular social media sites (e.g. Facebook). All interviews will be conducted through the HIPAA video-conferencing platforms, VSee and Zoom.

Specific Aims:

Phases I and II: To develop and refine a developmentally appropriate relationship skills session as an addition to the current CHTC intervention for 15-19 year old YMSM and their partners.

Phase III: To conduct a randomized controlled trial (RCT) comparing the efficacy of the adapted intervention for 15-24 year old YMSM versus a control condition, which is CTR or CHTC alone.

ELIGIBILITY:
Inclusion Criteria:

* Ages 15 to 24 years (inclusive) at time of screening
* Current U.S. resident
* Sufficient age for sexual consent in the current state of residence (assessed at both the individual and dyadic level)
* Self-identify that they are in an emotional and sexual relationship with another male
* Cisgender men (assigned male sex at birth and currently identifies as male) OR transgender men (assigned female at birth and identifies as male or transgender man
* Self-reports that they engaged in any kind of sexual activity (oral, vaginal, anal) in their lifetime
* Has access to computer/personal device/smart phone with internet access
* Self-report being HIV negative or unknown serostatus
* Speak and read English

Exclusion Criteria:

* Younger than age for consent without parental permission in the current state of residence
* Assigned female sex at birth and currently identifies as something other than male or transgender man
* Assigned male sex at birth but identifies as gender other than male or transgender man
* Aged 14 years or younger or 25 or older at the time of screening
* HIV-positive
* Not currently in an emotional and/or sexual relationship with another male
* Does not speak or read English
* Reports intimate partner violence in the past 6 months

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender men (assigned male sex at birth and currently identifies as male) OR transgender men (assigned female at birth and identifies as male or transgender man
Enrollment: 318 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Stephenson, PhD, Principal Investigator — University of Michigan; Kristi Gamarel, PhD, Principal Investigator — University of Michigan
Locations (1):
- Center for Sexuality and Health Disparities, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gamarel KE, Darbes LA, Hightow-Weidman L, Sullivan P, Stephenson R. The Development and Testing of a Relationship Skills Intervention to Improve HIV Prevention Uptake Among Young Gay, Bisexual, and Other Men Who Have Sex With Men and Their Primary Partners (We Prevent): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jan 2;8(1):e10370. doi: 10.2196/10370. PMID 30602433

RESULTS

PARTICIPANT FLOW:
Period: 3-Month Follow Up
Arm/Group | Control | Intervention
Started | 160 | 158
Completed | 121 | 120
Not Completed | 39 | 38
Not completed — Lost to Follow-up | 39 | 38
Period: 6-Month Follow Up
Arm/Group | Control | Intervention
Started | 160 | 158
Completed | 114 | 116
Not Completed | 46 | 42
Not completed — Lost to Follow-up | 46 | 42
Period: 9-Month Follow Up
Arm/Group | Control | Intervention
Started | 160 | 158
Completed | 116 | 115
Not Completed | 44 | 43
Not completed — Lost to Follow-up | 44 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 160 | 158 | 318
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 21 | 43
  Between 18 and 65 years | 138 | 137 | 275
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 21 [15 to 24] | 21 [15 to 24] | 21 [15 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 160 | 158 | 318
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 23 | 50
  Not Hispanic or Latino | 133 | 135 | 268
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 89 | 95 | 184
  More than one race | 33 | 27 | 60
  Unknown or Not Reported | 27 | 23 | 50
Region of Enrollment [Number; unit: participants]
  United States | 160 | 158 | 318
Sexual Risk Behavior [Count of Participants; unit: Participants] | 6 | 1 | 7
HIV Communication [Mean (Standard Deviation); unit: units on a scale] — Participants completed the 9-item Couples Efficacy to Reduce HIV Threat scale (Salazar, Stephenson, Sullivan, & Tarver, 2013). Participants responded to each item on 5-point Likert scale ranging from (1) strongly disagree to (5) strongly agree. The items were mean centered such that higher scores indicate that participants perceive that they can effectively communicate with their partner about HIV prevention strategies (range 1 to 5; sample α = 0.84).
  units on a scale | 4.5 (1.1) | 4.4 (0.9) | 4.5 (1.0)
PrEP use [Count of Participants; unit: Participants] | 14 | 7 | 21
HIV Testing [Count of Participants; unit: Participants] | 105 | 107 | 212
STI Testing [Count of Participants; unit: Participants] | 83 | 101 | 184

OUTCOME MEASURES:

1. Primary Outcome: Sexual Risk Behavior
Description: Anal or vaginal intercourse without condoms or PrEP that occurs with a person of known positive or unknown serostatus during follow-up period.
Time Frame: The number of participants who report sexual risk behavior at 3 months.
Population: Self-report of participants who reported sexual risk behavior.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 121 | 120
Participants | 1 | 2

2. Primary Outcome: Sexual Risk Behavior
Description: as for outcome 1
Time Frame: The number of participants who report sexual risk behavior at 6 months.
Population: Self-report of participants who reported sexual risk behavior.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 114 | 116
Participants | 0 | 2

3. Primary Outcome: Sexual Risk Behavior
Description: as for outcome 1
Time Frame: The number of participants who report sexual risk behavior at 9 months.
Population: Self-report of participants who reported sexual risk behavior.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 116 | 115
Participants | 0 | 1

4. Secondary Outcome: HIV Communication
Description: Participants completed the 9-item Couples Efficacy to Reduce HIV Threat scale .Participants responded to each item on 5-point Likert scale ranging from (1) strongly disagree to (5) strongly agree. The items were mean centered such that higher scores indicate that participants perceive that they can effectively communicate with their partner about HIV prevention strategies (range 1 to 5).
Time Frame: Mean at 3 months
Population: Self-report to scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 101 | 97
score on a scale | 4.6 (1) | 4.6 (0.9)

5. Secondary Outcome: HIV Communication
Description: Participants completed the 9-item Couples Efficacy to Reduce HIV Threat scale. Participants responded to each item on 5-point Likert scale ranging from (1) strongly disagree to (5) strongly agree. The items were mean centered such that higher scores indicate that participants perceive that they can effectively communicate with their partner about HIV prevention strategies (range 1 to 5).
Time Frame: Mean at 6 months
Population: Self-report on a scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 88 | 89
score on a scale | 4.5 (0.8) | 4.9 (0.9)

6. Secondary Outcome: HIV Communication
Description: as for outcome 5
Time Frame: Mean at 9 months
Population: Self-report on a scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 86 | 77
score on a scale | 4.8 (0.8) | 5.0 (0.6)

7. Secondary Outcome: PrEP Use
Description: Current PrEP use, which a self-report measure of whether the participant is currently using PrEP (yes/no).
Time Frame: The number of participants at 3 months
Population: Self-report of participants who reported that they were currently taking PrEP.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 121 | 120
Participants | 6 | 6

8. Secondary Outcome: PrEP Use
Description: Current PrEP use, which a self-report measure of whether the participant is currently using PrEP (yes/no)
Time Frame: The number of participants at 6 months
Population: Self-report of participants who reported that they were currently taking PrEP.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 114 | 116
Participants | 9 | 6

9. Secondary Outcome: PrEP Use
Description: Current PrEP use, which a self-report measure of whether the participant is currently using PrEP (yes/no)
Time Frame: The number of participants at 9 months
Population: Self-report of participants who self-reported that they were currently taking PrEP.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 116 | 115
Participants | 14 | 10

10. Secondary Outcome: HIV Testing
Description: Self-reported HIV testing in the past 3 months
Time Frame: The number of participants at 3-months
Population: Self-report of participants who had an HIV test in the past 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 121 | 120
Participants | 73 | 70

11. Secondary Outcome: HIV Testing
Description: Self-reported HIV testing in the past 3 months
Time Frame: The number of participants at 6 months
Population: Self-report of participants who had an HIV test in the past 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 114 | 116
Participants | 33 | 35

12. Secondary Outcome: HIV Testing
Description: Self-reported HIV testing in the past 3 months
Time Frame: The number of participants at 9 months
Population: Self-report of participants who reported that they had an HIV test in the past 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 116 | 115
Participants | 43 | 42

13. Secondary Outcome: STI Testing
Description: Any self-reported STI testing in the past 3 months
Time Frame: The number of participants at 3 months
Population: Self-report of participants who reported that they had an STI test in the past 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 121 | 120
Participants | 32 | 27

14. Secondary Outcome: STI Testing
Description: Any self-reported STI testing in the past 3 months
Time Frame: The number of participants at 6 months
Population: Self-report of participants who had an STI test in the past 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 114 | 116
Participants | 20 | 24

15. Secondary Outcome: STI Testing
Description: Any self-reported STI testing in the past 3 months
Time Frame: The number of participants at 9 months
Population: Self-report of participants who reported that they had an STI test in the past 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 116 | 115
Participants | 28 | 35

ADVERSE EVENTS:
Time Frame: 9 months
Description: Systemic assessment, which included standard questionnaire and regular investigator assessment.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/158
Serious Adverse Events (participants affected / at risk) | 0/160 | 0/158
Other Adverse Events (participants affected / at risk) | 0/160 | 0/158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03551938/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03551938/SAP_001.pdf